CLINICAL TRIAL: NCT00002348
Title: Phase II Evaluation of Mitoguazone Dihydrochloride in Patients With Refractory or Relapsed Non-Hodgkin's Lymphoma Associated With Acquired Immunodeficiency Syndrome
Brief Title: A Study of Mitoguazone Dihydrochloride in Patients With AIDS-Related Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Purpose: Treatment
Other Study IDs: 241A; IDD-007
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 1996-03

CONDITIONS: Lymphoma, Non-Hodgkin; HIV Infections
Keywords: Lymphoma, Non-Hodgkin; Acquired Immunodeficiency Syndrome; Lymphoma, AIDS-Related; Mitoguazone
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; HIV Infections; Acquired Immunodeficiency Syndrome; Lymphoma, AIDS-Related | interventions — Mitoguazone

INTERVENTIONS:
Drug: Mitoguazone

SUMMARY:
To estimate the response rate, response duration, clinical benefit, and toxicity of mitoguazone dihydrochloride (MGBG) in patients with AIDS-related refractory or relapsing non-Hodgkin's lymphoma (NHL).

DETAILED DESCRIPTION:
Patients receive infusions of MGBG on days 1 and 8 and every 2 weeks thereafter. It is suggested that a lumbar puncture be performed to evaluate for leptomeningeal disease.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV positivity by ELISA confirmed by Western blot.
* AIDS-related NHL that is refractory or relapsed.
* Life expectancy of at least 12 weeks.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Concomitant malignancy OTHER THAN curatively treated carcinoma in situ of the cervix; basal or squamous cell carcinoma of the skin; or non-active, non-visceral Kaposi's sarcoma not requiring active chemotherapy.
* Active uncontrolled bacterial infection, viral infection (other than herpes simplex), or fungal infection (other than oropharyngeal candidiasis) that requires treatment within 2 weeks of study entry.
* Significant cardiovascular disease.

Concurrent Medication:

Excluded:

* Hormonal therapy (except medications given for muscle wasting, such as testosterone or Megace).
* Other chemotherapy.
* Investigational anti-cancer drugs.

Concurrent Treatment:

Excluded:

* Concomitant radiation to sites other than CNS.

Patients with the following prior conditions are excluded:

Prior malignancy OTHER THAN curatively treated carcinoma in situ of the cervix; basal or squamous cell carcinoma of the skin; or non-active, non-visceral Kaposi's sarcoma not requiring active chemotherapy.

Recommended:

* Prophylaxis for PCP and oral candidiasis.

Required in patients with leptomeningeal disease:

* Intrathecal methotrexate or cytarabine (Ara-C).
* Leucovorin.

Required in patients with leptomeningeal disease:

Cranial radiation to a helmet field.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- ILEX Oncology Inc, San Antonio, Texas, United States

REFERENCES:
- [Background] Levine AM, Tulpule A, Tessman D, Kaplan L, Giles F, Luskey BD, Scadden DT, Northfelt DW, Silverberg I, Wernz J, Espina B, Von Hoff D. Mitoguazone therapy in patients with refractory or relapsed AIDS-related lymphoma: results from a multicenter phase II trial. J Clin Oncol. 1997 Mar;15(3):1094-103. doi: 10.1200/JCO.1997.15.3.1094. PMID 9060550